CLINICAL TRIAL: NCT04325802
Title: Treatment of Chronic Itch in Atopic Dermatitis With Opioid Antagonist Naltrexone and Effects on Skin Circadian Rhythm
Brief Title: Treatment of Chronic Itch in Atopic Dermatitis With Opioid Antagonist Naltrexone
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid-19 pandemic
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DERM-2019-28471
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis; Pruritus; Pruritus Chronic; Dermatitis
Keywords: Chronic Itch
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus; Dermatitis | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Placebo, then Intervention (Experimental): Patients will start with placebo in week 1 and cross over to Naltrexone in week 3. There will be a wash-out phase during week 2 using only moisturizer regularly and if necessary as rescue medications topical corticosteroids and/or antihistamines. The same rescue medications can be used during the following weeks of the cross-over treatment. At visit 2 and 4 patients will be asked the area where they are experiencing most intense itch and we will take there suction blisters (preferably on the trunk). Suction blisters will be taken after week 1 (1 week on treatment arm 1) and after week 3 (1 week on treatment arm 2).
  Interventions: Drug: Naltrexone; Other: Placebo
- Cohort 2: Intevention, then Placebo (Active Comparator): Patients will start with Naltrexone in week 1 and cross over to the palcebo treatment in week 3. There will be a wash-out phase during week 2 using only moisturizer regularly and if necessary as rescue medications topical corticosteroids and/or antihistamines. The same rescue medications can be used during the following weeks of the cross-over treatment. At visit 2 and 4 patients will be asked the area where they are experiencing most intense itch and we will take there suction blisters (preferably on the trunk). Suction blisters will be taken after week 1 (1 week on treatment arm 1) and after week 3 (1 week on treatment arm 2).
  Interventions: Drug: Naltrexone; Other: Placebo
- Circadian Rhythm of Itch (No Intervention): Patients in this arm will receive no intervention, only data collection.

INTERVENTIONS:
Drug: Naltrexone — 50mg Naltrexone daily
  Arms: Cohort 1: Placebo, then Intervention; Cohort 2: Intevention, then Placebo
Other: Placebo — Placebo (Mannitol) daily
  Arms: Cohort 1: Placebo, then Intervention; Cohort 2: Intevention, then Placebo

SUMMARY:
Purpose: To study the etiology and the epigenetic pathways leading to and regulating chronic itch. Similarly, to examine the mechanisms underlying skin changes, including epigenetic alterations while also testing the efficacy of opioid antagonists in atopic dermatitis. In this study, the investigators aim to examine chronic sensory disorder mechanisms related to chronic itch.

DETAILED DESCRIPTION:
Specific aims:

A1 Evaluate the underlying mechanism of itch severity in terms of circadian rhythm by collecting epidermis at different circadian stages using suction blisters. This will be done in AD patients with chronic itch. The cells will be isolated from part of the suction blisters and used to isolate and sequence RNA to evaluate and compare the differential protein and RNA expression in suction blister taken from symptomatic & non-symptomatic areas in patients with AD at different time points. The investigators will then correlate the itch severity symptoms to clock gene and opioid receptor levels and RNA expression differential pattern. A1 will be evaluated by study arm A and the results from this study will serve to decide on time point taking the suction blisters for the therapeutic/mechanistic studies (arm B and C).

A2 Investigate the mechanistic role and therapeutic efficacy of opioid receptors in chronic itch. For this purpose, a cross-over, placebo-controlled design will be used to treat patients with opioid receptor antagonist (Naltrexone) by expanding on our existing trial. The investigators will collect, evaluate, quantify and compare the differential protein and RNA expression in epidermis taken by suction blisters from symptomatic and non-symptomatic areas in patients with AD on Placebo or Naltrexone treatment. Transcriptome analysis will be focused, but not restricted to, analysis of neuroinflammatory and neuronal markers (including cytokines, GPCR and opioid receptors). Confirmation will occur using in-situ hybridization of biopsies to correlate specific cell type and location and qPCR expression of in vitro cultures. The binding studies using fluorescent labeled opioid ligands and internalization pattern will be carried out.

A3 Test the underlying mechanisms of the opioid system with nerve-keratinocyte interaction and possible effects on itch transduction from skin to nerves by using an in vitro neuron-keratinocyte co-culture model. Moreover, the investigators plan to validate itch-causing networks and pathways found in A2 using this in vitro model and will be able to evaluate calcium flux threshold changes after exposure to external stimuli (e.g. light, or mechanic stimuli) onto keratinocytes and neuronal somata under different opioid exposure conditions. The FC derived sensory neurons will be co-cultured with different patient KC. The investigators will test the reaction pattern of KC and transmission of the signal to connected peripheral sensory neurons by Fluo-4 AM Calcium imaging and electrophysiology. The reaction will be responding to the odorant Sandalore, as the investigators have previously published that Sandalore induces these desired calcium fluxes.

Apply the in vitro epithelial/nerve model to validate possible itch pathways identified by epigenetic analysis in the clinical trials by confirming the expression pattern with qPCR and functional assays on cells with CRISPR knockout of the RNA targets, opioid trafficking, calcium imaging and electrophysiology. Finally, further develop co-cultures between human skin and iPS-derived human peripheral neurons to perform functional studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD via simplified UK Working Group Criteria and a baseline PSGA score of 2 or greater
* Willingness to adhere to study protocol
* Subjects taking hormone-containing medications must be on a stable dose for 6 months prior to study start to avoid any confounding influence on sensory and pain perception

Exclusion Criteria:

* Use of topical or oral anti-inflammatory medications for 2 weeks prior to the study start.
* Use of topical or oral anti-histamines for 2 weeks prior to the study start (as rescue medication allowed).
* Use of topical or oral anti-pruritic agents for 2 weeks prior to the study start.
* Use of oral neuromodulatory agents for 2 months prior to study start.
* Current use of chronic pain medications (including opioids, antidepressants and anti-epileptic drugs).
* Use of nicotine-containing products for the past 6 months prior to study start.
* History of radiation or chemotherapy.
* History of traumatic injury on prospective test sites.
* Unstable thyroid function within the past 6 months prior to study start to exclude thyroid-related neuropathy
* Known history of central or peripheral nervous system dysfunction.
* History of acute hepatitis, chronic liver disease or end stage liver disease.
* History of human immunodeficiency virus (HIV) or acquired immune deficiency syndrome.
* History of neuropathy associated with chronic obstructive pulmonary disease, diabetes mellitus, documented exposure to organophosphates or heavy metals or polychlorinated biphenyls.
* Known nutritional deficiency (vitamin B12, vitamin D, iron or zinc) within 3 months prior to the study start.
* Use of illicit drugs within the past 6 months prior to study start and/or opioid use disorder.
* Regular use of opioids for chronic pain
* Lyme disease, porphyria, rheumatoid arthritis, Hansen's disease (leprosy) or use of antineoplastic chemotherapeutic agents.
* Subject has any medical condition that, in the judgment of the Investigator, would jeopardize the subject's safety following exposure to the administered medications.
* Adults lacking capacity to consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in Itch Intensity (Visual Analog Scale) | 1 week
  Change in itch intensity will be measured using a Visual Analogue scale (VAS). Scores range from 0 to 10, with higher scores indicating greater itch intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bigliardi, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided